CLINICAL TRIAL: NCT00700349
Title: Evaluation of Impacts of Access to Credit and Loan Size for Microcredit Clients in South Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovations for Poverty Action (Other)
Collaborators: Broadening Access and Strengthening Input Market Systems/USAID (Unknown); U.S. National Science Foundation (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other); Princeton University (Other); Social Science Research Council Program in Applied Economics (Unknown); Federal Reserve Bank of New York (Unknown)
Responsible Party: Dean Karlan, Innovations for Poverty Action
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: IPA-2004-SA
Record Dates: First submitted 2008-06-16; First posted 2008-06-18 (Estimated); Last update posted 2008-06-18 (Estimated); Status verified 2008-06

CONDITIONS: Mental Health; Depression; Stress
Keywords: depression; stress; microcredit; poverty; South Africa
MeSH Terms: conditions — Psychological Well-Being; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (No Intervention): Individuals who were rejected from receiving a loan from a micro-lending organization were randomized to continue receiving no loan.
- 2 (Experimental): Individuals who were rejected from receiving a loan from a micro-lending organization were randomized to receive a "second look," to be reconsidered for a loan by loan officers.
  Interventions: Other: Small loan

INTERVENTIONS:
Other: Small loan — Applicants in the treatment group were offered an interest rate, loan size, and maturity per the lender's standard underwriting criteria, involving a 4-month maturity at 11.75% per month, charged on the original balance (200% annual percentage rate).
  Arms: 2

SUMMARY:
This study involves randomization of individuals who were initially rejected from a micro-lending organization in South Africa. Subjects were placed into two arms: (1) not receiving a loan; (2) being reconsidered for a "second look." Of those in the second arm, 53% were then selected by the organization's loan officers to receive a standard loan for first-time borrowers. Mental health and financial data were collected at one timepoint: approximately 6-12 months after the subjects first applied for the loan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects were recruited from those who had been rejected from a lending organization for non-fraudulent or non-overindebtness reasons.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2004-09; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D), a 20-item questionnaire (0 = no risk, 60 = highest risk) | At follow-up (6-12 months after subject enrollment)
Perceived stress, measured using the Cohen's Perceived Stress Scale (PSS), a 10-item questionnaire (0 = no stress, 40 = high stress) | At follow-up (6-12 months after subject enrollment)

SECONDARY OUTCOMES:
Household income, measured by a variety of questions that asked about all sources of income obtained by all members of the applicant's household. | At follow-up (6-12 months after subject enrollment)

CONTACTS AND LOCATIONS:
Overall Officials: Dean Karlan, PhD, Principal Investigator — Innovations for Poverty Action; Jonathan Zinman, PhD, Principal Investigator — Dartmouth University; Lia Fernald, PhD, Principal Investigator — University of California, Berkeley
Locations (3):
- South Africa (3):
  - Innovations for Poverty Action, Cape Town
  - Innovations for Poverty Action, Durban
  - Innovations for Poverty Action, Port Elizabeth